CLINICAL TRIAL: NCT02928770
Title: A Disposable Device NAS to Treat Obstructive Sleep Apnea and Snoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Seven Dreamers Laboratories (Unknown)
Responsible Party: Principal Investigator, Clete A. Kushida, Medical Director/Clinic Chief, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 32492
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-12

CONDITIONS: Obstructive Sleep Apnea; Snoring
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Nastent (Experimental): A baseline sleep study is obtained from the subject, without wearing the device. The individual wears the device at home for at least 7 nights, and then returns to the sleep lab for an in-laboratory sleep study while wearing the device.
  Interventions: Device: Nastent

INTERVENTIONS:
Device: Nastent — Use of the device while at home and in the sleep lab

SUMMARY:
The purpose of this research study is to test a new approach for treating patients with obstructive sleep apnea and/or snoring. The new nasal device, nastent (NAS: nasal airway stent), appears to be a useful alternative or additive treatment.

DETAILED DESCRIPTION:
The nasal stent basically helps to splint the soft palate open. Subjects have a baseline (diagnostic) sleep study without wearing the device. Subjects are then fitted with the device and then subjects wear the device for at least 7 nights during their sleep while at home. Subjects then return for a repeat in-laboratory sleep study while wearing the device. The primary outcome is to assess the effectiveness of the device by change in the apnea-hypopnea index (number of sleep-related abnormal breathing events per hour of sleep) while wearing the device compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Adults that are 18 years of age or older who had a prior sleep-study within the past 6 months that confirmed a diagnosis of obstructive sleep apnea, and with body mass index less than 30 kg/m2.

Exclusion Criteria:

* Children, pregnant women, homeless, economically disadvantaged individuals, and those who are unable to comprehend or understand English, or follow instructions were excluded. Persons with body mass index equal or greater than 30 kg/m2 were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-02; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clete A Kushida, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Sleep Medicine, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nastent
Started | 32
Completed | 30
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Nastent
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 18
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 30
Apnea-Hypopnea Index [Mean (Standard Deviation); unit: events/hour] — Abnormal breathing events (apneas = complete pauses in oronasal airflow; hypopneas = decreases in oronasal airflow) per hour of sleep. This is measured through polysomnography (sleep study) by a nasal thermistor and oral pressure sensor.
  events/hour | 34.9 (23.8)

OUTCOME MEASURES:

1. Primary Outcome: Apnea-Hypopnea Index (AHI)
Description: Abnormal breathing events (apneas = complete pauses in oronasal airflow; hypopneas = decreases in oronasal airflow) per hour of sleep. This is measured through polysomnography (sleep study) by a nasal thermistor and oral pressure sensor.
Time Frame: In-lab sleep study obtained at least 7 nights following use of the device at home
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Nastent
Number analyzed (Participants) | 30
events/hour | 30.0 (20.3)
Statistical Analysis 1: Comparison: Nastent; Test type: Other; p = 0.0559, t-test, 2 sided; Comparison between baseline and experimental (Nastent) conditions

ADVERSE EVENTS:
Time Frame: 7.5 months (baseline visit to end-of-study visit)
Arm/Group | Nastent
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT02928770/Prot_000.pdf
  • Statistical Analysis Plan (2014-12-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT02928770/SAP_001.pdf